CLINICAL TRIAL: NCT05276037
Title: Extension of Liver Transplantation Opportunity to Patients Suffering From Milan-out, Up-to-7-in, Hepatocellular Carcinoma: a Prospective Belgian Study of the Value of Negative 18FDG PET/CT
Brief Title: Value of Negative 18FDG PET/CT in Milan Out, Up-to-seven in, HCC Transplant Candidates
Status: Recruiting | Type: Observational
Sponsor: University of Liege (Other)
Collaborators: University Hospital, Ghent (Other); Free University of Brussels (Other); University Hospital, Antwerp (Other); Universitaire Ziekenhuizen KU Leuven (Other); Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Principal Investigator, Olivier Detry MD PhD, Associate professor, Surgical head of the liver transplantation program, University of Liege
Other Study IDs: B707201939900
Record Dates: First submitted 2022-03-02; First posted 2022-03-11 (Actual); Last update posted 2022-09-01 (Actual); Status verified 2022-08

CONDITIONS: Hepatocellular Carcinoma
Keywords: Liver transplantation; Milan criteria; Prognostic factor; PET CT; recurrence
MeSH Terms: conditions — Carcinoma, Hepatocellular; Recurrence | interventions — Liver Transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples Without DNA — The HCC liver explant stored in the local biobank of the transplant center.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study group: Milan-out, up-to-7-in, PET negative (≤1.15) HCC patients
  Interventions: Other: Liver transplantation
- Control group: Milan-in HCC patients
  Interventions: Other: Liver transplantation

INTERVENTIONS:
Other: Liver transplantation — Both groups will receive the same advantages on the LT waiting list (SE points)

SUMMARY:
Hepatocellular carcinoma (HCC) is a rising public health concern with few curative options but liver transplantion (LT) in highly selected cases. LT could save many other HCC patients but organ shortage has lead to the necessity of selection of patients with the best survival chances, namely the Milan criteria. Hepatocellular carcinoma (HCC) is the fifth most common cancer, and the third cause of cancer related-death worldwide. HCC incidence is rising in Western countries including Belgium. There are more than 1,000 new HCC diagnoses in Belgium every year, but only 90 to 100 patients suffering from HCC are listed for liver transplantation (LT). In fact, the scarcity of organ donors has forced the development of strict criteria to limit LT to patients who are likely to have excellent outcomes. The universally accepted LT criteria for HCC are the Milan criteria (1 HCC nodule ≤5 cm or 3 nodules ≤3cm) that lead to a low rate of post-LT recurrence (>80% of disease free recurrence at 5 years). The majority of patients suffering from HCC outside the Milan criteria at the time of diagnosis is not eligible for LT and is therefore limited to palliative care. It is however considered that some of these patients with HCC outside the Milan criteria may benefit from LT with an acceptable risk of recurrence and chances of long-term disease-free survival (DFS). This fact has led to the extension of LT criteria for HCC in some centres in different countries, as for example the University of California San Francisco (UCSF) criteria, the up-to-seven criteria or the Asan criteria.

The Belgian Liver-Intestine Allocation Committee (Be-LIAC) is a section of the Belgian Transplantation Society (BTS) composed of the 6 LT Belgian centres in charge of coordinating deceased LT activity in Belgium with the help of Eurotransplant. Be-LIAC has already built a retrospective HCC database that was successfully used for several scientific studies allowing international presentations and publications. Based on this successful experience, Be-LIAC is keen to continue with this national collaboration to initiate a prospective clinical observational database to better study the results of LT in Belgium and to evaluate potential of extension of LT criteria in HCC patients. Inclusion in this database will not change patient management or the allocation process of the liver grafts in Belgium. This project is financed by a 4-year (2019-2022) grant of the Belgian "Fondation contre le cancer" / "Stichting tegen Kanker".

DETAILED DESCRIPTION:
All adult patients (> 18 and < 80 years) suffering from HCC and discussed for potential deceased or living related LT during multidisciplinary oncologic meetings in the 6 Belgian LT centres will be consecutively included in the prospective database after signing an informed consent form. Date of inclusion will be the date of discussion at the first multidisciplinary oncological meeting. All patients who are not contra indicated for LT due to general medical conditions (as presented in the exclusion criteria) or due to HCC staging (evidence of extrahepatic extension or cancerous macroscopic invasion of a liver vein at imaging) will be included in the database. These patients will be either directly listed on the Eurotransplant waiting list if considered within the local LT criteria by the given centre, or potentially listed after successful down-staging or HCC recurrence after a first attempt of curative management (ex: resection, radiofrequency ablation (RFA), ….).

A prospective, secured, anonymized (GDPR compliant), web-based database will be constructed with the help of an experienced company.

For LT listing, diagnosis of HCC will be based on international recommendations and Eurotransplant rules, either on biopsy or on imaging (AFP >400 ng/mL and 1 positive result with hypervascularisation on CT and/or MRI), or AFP < 400ng/mL and 2 positive results with CT and MRI). Hepatic lesions of <1cm will not be considered for preoperative radiologic staging. All of the relevant liver images will be stored in a secured (GDPR compliant) web-based server and will be reviewed by a multicentre panel of expert radiologists in order to confirm the radiologic staging according to Milan and up-to-seven criteria.

Registration of HCC patients on the Eurotransplant waiting list will not be modified. Transplant candidates will be registered on the LT waiting list according to Eurotransplant and Be-LIAC allocation rules:

* 1 HCC nodule > 2cm: labMELD score;
* HCC within the Milan criteria: (1 HCC nodule ≤ 5 cm or 3 nodules ≤ 3cm) exceptional standard exception (SE) MELD points;
* HCC outside the Milan criteria but successfully down-staged to inside Milan criteria: exceptional SE MELD points;
* HCC outside Milan criteria, within up-to-7 criteria, PET negative (≤ 1.15): exceptional SE MELD points;
* HCC outside Milan criteria, within up-to-7 criteria, PET positive (> 1.15) or outside up-to-7 criteria: labMELD score.

Nodules ≤ 1 cm will be taken into account.

After transplantation, patients will undergo regular life-long immunosuppression according to the centre preferences. In the context of a malignant disease, the use of mTOR inhibitors will be encouraged but not mandatory, as suggested in the recent literature. The type of immunosuppression (induction therapy, calcineurin inhibitors, mTOR inhibitors, antimetabolites, steroids) will be recorded in the database. No adjuvant therapy will be performed in patients without evidence of recurrence.

Posttransplant tumour surveillance program will be standard for LT recipients with HCC and will consist in at least whole body CT every 6 months during the first 2 years, and AFP level measurement every 3-6 months during the entire follow-up period in patients with elevated pretransplant AFP. The date and site of recurrence will be recorded as well as survival data. Management of recurrence will be performed according to the centre policy and recorded in the database. As for other solid organ transplant recipients, all LT patients included in this study will be indefinitely followed by local transplant centres, allowing mid- and long-term (10 years) follow-ups.

Recorded data

* Patient's characteristics: Patient code generated by Eonix, internal patient code at the transplant center, Eurotransplant listing with the number and date of registration, ET listing criteria, country of residence, ethnicity, age, gender, blood group, BMI, viral status, cause of cirrhosis, diabetic status, smoking status, cancer status, history of liver and/or obesity surgery, cause of chronic liver disease, ascites and encephalopathy grade and Milan status at the Eurotransplant listing. If an HCC would have been treated in the past, more information will be required.
* HCC Data: - CT scan with the date, number of nodules and their sizes as well as their classification (TNM grade according to UICC 2018);

  - MRI with the date, the numbers of nodules and their size and their classification (TNM grade); - tumour biopsy with date and characteristics (differentiation, invasion) if performed; - FDG-PET / CT with the characteristics SUV max (> 1.15) or SUV max (≤1.15); Medium SUV; the ratio between max SUV of the tumour with max SUV of a "normal" liver .
* Pre-transplant visits every 3 months: date, hemoglobin, platelets, white cells, neutrophils, lymphocytes, monocytes, international normalized ratio (INR), total bilirubin, creatinin, C-reactive protein (CRP), AFP, CA19-9, albumin and natrium. Lab-MELD score, encephalopathy and ascites grade, allowing determining Child Pugh score, CT scan/MRI every 3 to 4 months to monitor the nodules and their evolution. In addition, in some patients, blood samples will be stored in the biobank center. Additional informed consent will need to be signed by the patient to allow to retain vital biological data for future research. Standard neo-adjuvant HCC management (also called "bridge-to-transplant") will be performed according to the local multidisciplinary team decision, including resection, RFA, chemoembolization, radioembolization, Sorafenib, stereotaxic radiotherapy or no therapy. These informations will be included in the database. While on the LT waiting list, patients will be followed by CT/MRI and AFP level every 3 to 4 months, allowing the evaluation of the evolution of the tumour size and the ΔAFP. Response to neo-adjuvant therapy will be determined according to the modified Response Evaluation Criteria in Solid Tumors (mRECIST): complete-response (CR), partial-response (PR), stable-disease (SD) and progressive-disease (PD).
* Liver transplant data: Recipients pretransplant last lab values: hemoglobin, platelets, white cells, neutrophils, lymphocytes, monocytes, INR, total bilirubin, creatinine, CRP, AFP, albumin, natrium, encephalopathy and ascites grade, waiting time before transplant, lab and exceptional MELD score at LT, Eurotransplant donor number, age of donor, type of donor, type of graft, graft origin, donor total bilirubin, ET donor risk index (ET-DRI), graft biopsy, time of ischemia, blood transfusion during surgery and after, need renal support, transaminase peak, total bilirubin at day 7, number of days in ICU, number of hospitalisation days.
* Pathology of explanted livers. Number of nodules and their sizes as well as their classification (TNM grade according to UICC 2018). These samples will be stored in the center's biobank to allow for further analyses needed for research in liver oncology. A consent must be signed by the patient.
* Follow up visits after LT: 1 month, 3 months, 6 months, 9 months, 12 months, 15 months, 18 months, 21 months, 24 months, 30 months, 36 months, 42 months, 48 months, 54 months, 60 months, 66 months, 72 months, 78 months, 84 months, 90 months, 96 months, 102 months, 108 months, 114 months, 120 months:

Biology at follow up: AFP, tacrolimus level, everolimus level. Recorded informations: immunosuppression, graft survival, cause of transplant failure, the date of retransplantation, cause of patient death, recurrence of HCC and its location and planned treatment. A body CT will be performed at 6 months, 12 months, 18 months, 24 months, 32 months, 44 months and 60 months.

ELIGIBILITY:
Inclusion Criteria:

* HepatoCellular Carcinoma
* Liver transplant candidate after multidisciplinary disccuss

Exclusion Criteria:

* Patients < 18y or > 80yr old
* Patients considered contra-indicated (CI) for LT due to non-liver-related medical problems (age, other cancer, psychiatric disease, uncontrolled infection, no compliance, active alcohol abuse, cardiac CI, pulmonary CI, surgical CI, other medical CI);
* Patients contra-indicated for LT due to the HCC: extra-hepatic metastases (M+), lymphatic involvement (N+), macro-vascular invasion.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients (> 18 and < 80 years) suffering from HCC and discussed for potential deceased or living related LT (including combined transplantation) during multidisciplinary oncology meetings in the 6 Belgian LT centres (either direct listing for LT on the Eurotransplant waiting list or potential listing after downstaging or recurrence after other treatment).
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2029-01-01 (Estimated)

PRIMARY OUTCOMES:
Survival | 1,2, 5, and 10 years after LT
  Intention-to-treat (at LT waiting list registration) and post LT disease-free (DFS), recurrence-free (RFS) and overall survivals (OS)

SECONDARY OUTCOMES:
FDG PET-CT as a pronostic factor for HCC patients undergoing liver transplantation | 1,2, 5, and 10 years after LT
  Comparison of FDG-PET/CT to the other prognostic HCC prognostic factors, as the radiologic and pathologic Milan criteria, the UCSF criteria, the up-to-seven criteria, the Asan criteria and the AFP model
FDG PET-CT value in Milan-in patients | 1,2, 5, and 10 years after LT
  Evaluation of the value of positive or negative FDG-PET/CT in Milan-in HCC patients listed for LT and the impact on outcome in these patients

CONTACTS AND LOCATIONS:
Locations (6):
- Belgium (6):
  - University Hospital, Antwerp, Antwerp
  - Free University of Brussels, Brussels
  - University Hospital, Ghent, Ghent
  - Catholic University of Louvain, Leuven
  - Leuven University hospital, Leuven
  - ULiège, Liège

IPD SHARING:
Plan to Share IPD: No